CLINICAL TRIAL: NCT00002004
Title: A Phase I Study of the Safety and Pharmacokinetics of Recombinant CD4 (rCD4) in Patients With AIDS and AIDS-Related Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 064A; CO030g; Serial Number 002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — CD4 Antigens

INTERVENTIONS:
Drug: CD4 Antigens

SUMMARY:
To determine the safety profile and maximum tolerated dose (MTD) of recombinant soluble human CD4 (rCD4) therapy in patients with AIDS or AIDS related complex (ARC). To assess pharmacokinetic properties of rCD4 in humans. To obtain a preliminary indication of the antiviral effects of rCD4 in patients with AIDS and AIDS related complex (ARC).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositivity.
* Diagnosis of AIDS or AIDS related complex (ARC).
* Failure to tolerate or respond to zidovudine (AZT) or decided to decline AZT therapy.
* The ability to sign a written informed consent form prior to treatment.
* A willingness to abstain from all other experimental therapy for HIV infection during the entire study period.
* A life expectancy of at least 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Serious active opportunistic infections.
* Malignancies other than Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Corticosteroids.
* Nonsteroidal anti-inflammatory agents (NSAI).
* Other experimental therapy.

Patients with the following are excluded:

* Serious active opportunistic infections.
* Malignancies other than Kaposi's sarcoma.

Prior Medication:

Excluded within 3 weeks of study entry:

* Zidovudine (AZT).
* Chemotherapy.
* Immunomodulators.
* Other experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Genentech Inc, South San Francisco, California, United States